CLINICAL TRIAL: NCT04454918
Title: A Phase 1 Study to Assess Absolute Bioavailability of TAK-906 and to Characterize Mass Balance, Pharmacokinetics, Metabolism, and Excretion of [14C]-TAK-906 in Healthy Male Subjects
Brief Title: Study to Assess Absolute Bioavailability (ABA) of TAK-906 and to Characterize Mass Balance, Pharmacokinetics (PK), Metabolism, and Excretion of [14C]-TAK-906 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-906-1007; U1111-1254-4588 (Other: WHO)
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Results first posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — trazpiroben

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-906 50 mg + [14C]-TAK-906 100 mcg + [14C]-TAK-906 50 mg (Experimental): TAK-906 50 mg, capsule, orally, once on Day 1, followed by [14C]-TAK-906 100 micrograms (μg) [approximately 1 microcurie (μCi)], IV infusion, once on Day 1 of Treatment Period 1, followed by a Washout Period of 7 days, further followed by [14C]-TAK-906 50 mg (approximately 100 μCi), solution, orally, once on Day 1 of Treatment Period 2.
  Interventions: Drug: TAK-906 Oral Capsule; Drug: [14C]-TAK-906 Intravenous Infusion; Drug: [14C]-TAK-906 Oral Solution

INTERVENTIONS:
Drug: TAK-906 Oral Capsule — TAK-906 capsule.
Drug: [14C]-TAK-906 Intravenous Infusion — [14C]-TAK-906 intravenous infusion.
Drug: [14C]-TAK-906 Oral Solution — [14C]-TAK-906 oral solution.

SUMMARY:
The purpose of this study is to determine ABA of TAK-906 following single oral (capsule) administration of 50 milligram (mg) of TAK-906 and single intravenous (IV) microtracer dose administration of 100 microgram (μg) (approximately 1 microcurie [μCi]) of [14C]-TAK-906 in Period 1 (ABA), and to determine the mass balance of TAK-906 in urine and feces following a single oral (solution) administration of 50 mg (approximately 100 μCi) of [14C]-TAK-906 in Period 2 (absorption, distribution, metabolism, and elimination [ADME]).

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-906. The study will determine ABA in Period 1, and ADME, and mass balance of TAK-906 after single oral administration in Period 2 in healthy adult male participants. Plasma and urine samples will be collected for PK determination; plasma, whole blood, urine, and feces samples will be collected for total radioactivity (TRA) determination; and plasma, urine, and feces samples will be collected to characterize the metabolite profiles of TAK-906.

The study will enroll approximately 6 participants. The study is designed to consist of 2 periods: Period 1 (ABA study period) and Period 2 (ADME study period). In Period 1 (ABA study period), all participants will receive single unlabeled oral 50 mg dose of TAK-906 as capsule followed by microdose of 100 μg (approximately 1 μCi) [14C]-TAK-906 as intravenous infusion followed by a washout period of at least 7 days before the dose in Period 2. In Period 2 (ADME study period), all participants will receive a single dose of 50 mg (approximately 100 μCi) [14C]-TAK-906 as an oral solution.

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 65 days including screening period. Participants will be contacted approximately 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study.
2. Body mass index (BMI) greater than or equal to (>=) 18.0 and less than (˂) 30.0 kilogram per square meter (kg/m^2) at screening.

Exclusion Criteria:

1. QT interval corrected for heart rate using Fridericia's formula (QTcF) interval is greater than (>) 450 millisecond (msec) or Electrocardiogram (ECG) findings are deemed abnormal with clinical significance by the Investigator or designee at screening.
2. Estimated creatinine clearance less than (<) 90 milliliter per minute (mL/min) at screening.
3. Has tattoo(s) or scarring at or near the site of intravenous (IV) infusion or any other condition which may interfere with infusion site examination, in the opinion of the Investigator.
4. Has infrequent bowel movements (less than approximately once per day) within 30 days prior to first dosing.
5. Has received radiolabeled substances or has been exposed to radiation sources within 12 months of first dosing or is likely to receive radiation exposure or radioisotopes within 12 months of last dosing such that participation in this study would increase their total exposure beyond the recommended levels considered safe (that is weighted annual limit recommended by the International Commission on Radiological Protection [ICRP] of 3000 milli roentgen equivalent man [mrem]).
6. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
7. Donation of blood or significant blood loss within 56 days prior to the first dosing.
8. Plasma donation within 7 days prior to the first dosing.
9. Unable to refrain from or anticipates the use of:

   * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing and throughout the study. Acetaminophen (up to 2 g per 24 hour period) and Milk of Magnesia® (that is, magnesium hydroxide [less than or equal to (<=) 60 mL per day after Day 3 in Period 1 and after Day 8 in Period 2]) may be permitted during the study, only after dosing, if necessary to treat adverse events (AEs). Additional administration of Milk of Magnesia® may be administered on other days at discretion of the Investigator.
   * Any drugs known to significantly affect the absorption, distribution, metabolism or elimination of TAK-906 within 28 days prior to the first dosing and throughout the study. Appropriate sources (example, Flockhart Table TM) will be consulted to confirm lack of PK/pharmacodynamics interaction with study drug.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 30 July 2020 to 29 September 2020.
Pre-assignment Details: Healthy male participants were enrolled in this study to receive TAK-906 capsule followed by radio-labelled TAK-906 intravenous (IV) infusion on Day 1 of Treatment Period 1 and radio-labelled TAK-906 oral solution on Day 1 of Treatment Period 2. There was a 7-day Washout Period between the two periods.
Groups:
- TAK-906 50 mg + [14C]-TAK-906 100 μg + [14C]-TAK-906 50 mg: TAK-906 50 mg, capsule, orally, once on Day 1, followed by [14C]-TAK-906 100 micrograms (μg) [approximately 1 microcurie (μCi)], IV infusion, once on Day 1 of Treatment Period 1, followed by a Washout Period of 7 days, further followed by [14C]-TAK-906 50 mg (approximately 100 μCi), solution, orally, once on Day 1 of Treatment Period 2.
Period: Treatment Period 1 (Day 1)
Arm/Group | TAK-906 50 mg + [14C]-TAK-906 100 μg + [14C]-TAK-906 50 mg
Started | 6
Completed | 6
Not Completed | 0
Period: Washout Period (Day 2 to 8)
Arm/Group | TAK-906 50 mg + [14C]-TAK-906 100 μg + [14C]-TAK-906 50 mg
Started | 6
Completed | 6
Not Completed | 0
Period: Treatment Period 2(Day9[Day1of Period2])
Arm/Group | TAK-906 50 mg + [14C]-TAK-906 100 μg + [14C]-TAK-906 50 mg
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who received at least one dose of the study drug.
Groups:
- TAK-906 50 mg + [14C]-TAK-906 100 μg + [14C]-TAK-906 50 mg: TAK-906 50 mg, capsule, orally, once on Day 1, followed by [14C]-TAK-906 100 μg (approximately 1 μCi), IV infusion, once on Day 1 of Treatment Period 1, followed by a Washout Period of 7 days, further followed by [14C]-TAK-906 50 mg (approximately 100 μCi), solution, orally, once on Day 1 of Treatment Period 2.
Arm/Group | TAK-906 50 mg + [14C]-TAK-906 100 μg + [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Weight [Mean (Standard Deviation); unit: kg] | 87.30 (13.242)
Height [Mean (Standard Deviation); unit: cm] | 181.7 (8.19)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = weight (kg)/height (m)^2
  kg/m^2 | 26.408 (2.9179)

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Absolute Bioavailability Based on Ratio of Dose Normalized Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC∞ ) for TAK-906
Description: Bioavailability is defined as the proportion of a drug which enters the circulation when introduced into the body and so is able to have an active effect. Percent absolute bioavailability for plasma TAK-906, calculated as geometric least squares mean ratio: [Actual Dose (IV) x AUC∞ (oral)] / [Actual Dose (oral) x AUC∞ (IV)] multiplied (x) 100, where AUC∞ for IV infusion was normalized to a 50 mg dose.
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 1
Population: Pharmacokinetic (PK) Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the oral dose of TAK-906 50 mg capsules followed by [14C]-TAK-906 100 μg [approximately 1 μCi], IV infusion in Period 1 were evaluated for this outcome measure.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: percent absolute bioavailability
Groups:
- TAK-906 50 mg + [14C]-TAK-906 100 μg: TAK-906 50 mg, capsule, orally, once on Day 1, followed by [14C]-TAK-906 100 μg [approximately 1 μCi], IV infusion, once on Day 1 of Treatment Period 1.
Arm/Group | TAK-906 50 mg + [14C]-TAK-906 100 μg
Number analyzed (Participants) | 6
percent absolute bioavailability | 9.12 [7.49 to 11.10]

2. Primary Outcome: Period 2: Cum%Dose (UR): Cumulative Percentage of Total Radioactivity Excreted in Urine for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose in Treatment Period 2
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the dose of [14C]TAK-906 50 mg oral solution in Treatment Period 2 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Groups:
- [14C]-TAK-906 50 mg: [14C]-TAK-906 50 mg (approximately 100 μCi), solution, orally, once on Day 1 of Treatment Period 2.
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
percentage of dose | 2.162 (21.8)

3. Primary Outcome: Period 2: Cum%Dose (FE): Cumulative Percentage of Total Radioactivity Excreted in Feces for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
percentage of dose | 94.44 (1.9)

4. Primary Outcome: Period 2: Combined Cum%Dose: Cumulative Combined Percent of Total Radioactivity Excreted in Urine and Feces for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
percentage of dose | 96.65 (1.7)

5. Secondary Outcome: Period 1: Cmax: Maximum Observed Plasma Concentration for TAK-906 and Metabolite (M23) After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the oral dose of TAK-906 50 mg capsules in Treatment Period 1 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- TAK-906 50 mg: TAK-906 50 mg, capsule, orally, once on Day 1 of Treatment Period 1.
Arm/Group | TAK-906 50 mg
Number analyzed (Participants) | 6
ng/mL
  TAK-906 | 29.72 (49.2)
  Metabolite (M23) | 2.293 (50.4)

6. Secondary Outcome: Period 1: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-906 and M23 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 1
Population: as for outcome 5
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | TAK-906 50 mg
Number analyzed (Participants) | 6
hour (hr)
  TAK-906 | 1.750 [1.00 to 4.00]
  Metabolite (M23) | 1.750 [1.00 to 4.00]

7. Secondary Outcome: Period 1: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-906 and M23 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | TAK-906 50 mg
Number analyzed (Participants) | 6
ng*hr/mL
  TAK-906 | 78.62 (24.5)
  Metabolite (M23) | 6.185 (37.3)

8. Secondary Outcome: Period 1: AUC%Extrap: Percent of Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC∞) Extrapolated for TAK-906 and M23 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the oral dose of TAK-906 50 mg capsules in Treatment Period 1 were evaluated for this outcome measure. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC
Arm/Group | TAK-906 50 mg
Number analyzed (Participants) | 6
percentage of AUC
  TAK-906 | 0.6598 (58.5)
  Metabolite (M23): number analyzed (Participants) | 5
  Metabolite (M23) | 4.288 (67.7)

9. Secondary Outcome: Period 1: t(1/2)z : Terminal Disposition Phase Half-life for TAK-906 and M23 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (hr)
Arm/Group | TAK-906 50 mg
Number analyzed (Participants) | 6
hours (hr)
  TAK-906 | 3.892 (73.1)
  Metabolite (M23): number analyzed (Participants) | 5
  Metabolite (M23) | 1.722 (24.1)

10. Secondary Outcome: Period 1: Vz/F: Apparent Volume of Distribution During the Terminal Elimination Phase for TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | TAK-906 50 mg
Number analyzed (Participants) | 6
Liters | 3545 (78.3)

11. Secondary Outcome: Period 1: CL/F: Apparent Total Plasma Clearance for TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | TAK-906 50 mg
Number analyzed (Participants) | 6
L/hr | 631.3 (24.2)

12. Secondary Outcome: Period 1: Ceoi: Plasma Total Radioactivity Concentration at the End of Infusion for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the [14C]-TAK-906 μg IV infusion in Treatment Period 1 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogramequivalents/milliliter(ng eq/mL)
Groups:
- [14C]-TAK-906 100 μg: [14C]-TAK-906 100 μg (approximately 1 μCi), IV infusion, once on Day 1 of Treatment Period 1, after the TAK-906 oral dose, followed by a Washout Period of 7 days.
Arm/Group | [14C]-TAK-906 100 μg
Number analyzed (Participants) | 6
nanogramequivalents/milliliter(ng eq/mL) | 3.529 (18.5)

13. Secondary Outcome: Period 1: AUClast: Area Under the Plasma Total Radioactivity Concentration-time Curve From Time 0 to Last Quantifiable Concentration for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]-TAK-906 100 μg
Number analyzed (Participants) | 6
ng eq*hr/mL | 2.047 (14.3)

14. Secondary Outcome: Period 1: AUC∞: Area Under the Plasma Total Radioactivity Concentration-time Curve From Time 0 to Infinity for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the [14C]-TAK-906 μg IV infusion in Treatment Period 1 were evaluated for this outcome measure. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]-TAK-906 100 μg
Number analyzed (Participants) | 3
ng eq*hr/mL | 1.976 (14.2)

15. Secondary Outcome: Period 1: t(1/2)z: Terminal Disposition Phase Half-life of Plasma Total Radioactivity Concentration for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | [14C]-TAK-906 100 μg
Number analyzed (Participants) | 3
hr | 10.847 (137.1)

16. Secondary Outcome: Period 1: Ceoi: Plasma Concentration at the End of Infusion for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms (pg)/mL
Arm/Group | [14C]-TAK-906 100 μg
Number analyzed (Participants) | 6
picograms (pg)/mL | 3795 (14.1)

17. Secondary Outcome: Period 1: CL: Total Clearance for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | [14C]-TAK-906 100 μg
Number analyzed (Participants) | 6
L/hr | 57.55 (11.8)

18. Secondary Outcome: Period 1: Vss: Volume of Distribution During the Terminal Disposition Phase for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | [14C]-TAK-906 100 μg
Number analyzed (Participants) | 6
Liters | 33.04 (14.2)

19. Secondary Outcome: Period 1: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to Last Quantifiable Concentration for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/mL
Arm/Group | [14C]-TAK-906 100 μg
Number analyzed (Participants) | 6
pg*hr/mL | 1549 (10.7)

20. Secondary Outcome: Period 1: AUC%Extrap: Percent of Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC∞) Extrapolated for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC
Arm/Group | [14C]-TAK-906 100 μg
Number analyzed (Participants) | 6
percentage of AUC | 0.3908 (42.6)

21. Secondary Outcome: Period 1: t(1/2)z: Terminal Disposition Phase Half-life for [14C]-TAK-906
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | [14C]-TAK-906 100 μg
Number analyzed (Participants) | 6
hr | 1.196 (21.2)

22. Secondary Outcome: Period 2: Cmax: Maximum Observed Plasma Concentration for TAK-906 and M23 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the dose of [14C]-TAK-906 50 mg oral solution in Treatment Period 2 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
ng/mL
  TAK-906 | 26.81 (31.1)
  Metabolite (M23) | 1.086 (48.1)

23. Secondary Outcome: Period 2: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-906 and M23 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 22
Measure: Median (Full Range); unit: hr
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
hr
  TAK-906 | 0.500 [0.50 to 1.50]
  Metabolite (M23) | 0.999 [0.50 to 1.50]

24. Secondary Outcome: Period 2: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-906 and M23 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
ng*hr/mL
  TAK-906 | 46.54 (23.5)
  Metabolite (M23) | 2.111 (47.7)

25. Secondary Outcome: Period 2: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-906 and M23 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the dose of [14C]-TAK-906 50 mg oral solution in Treatment Period 2 were evaluated for this outcome measure. Number analyzed is the number of participants with data available for analysis for the given category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
ng*hr/mL
  TAK-906 | 49.40 (18.6)
  Metabolite (M23): number analyzed (Participants) | 5
  Metabolite (M23) | 2.490 (50.1)

26. Secondary Outcome: Period 2: AUC%Extrap: Percent of Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC∞) Extrapolated for TAK-906 and M23 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
percentage of AUC
  TAK-906 | 3.993 (96.7)
  Metabolite (M23): number analyzed (Participants) | 5
  Metabolite (M23) | 8.013 (50.0)

27. Secondary Outcome: Period 2: t(1/2)z: Terminal Disposition Phase Half-life for TAK-906 and M23 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
hr
  TAK-906 | 9.993 (29.4)
  Metabolite (M23): number analyzed (Participants) | 5
  Metabolite (M23) | 1.833 (57.9)

28. Secondary Outcome: Period 2: Vz/F: Apparent Volume of Distribution During the Terminal Elimination Phase for TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
Liters | 14430 (29.7)

29. Secondary Outcome: Period 2: CL/F: Apparent Total Plasma Clearance for TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
L/hr | 1007 (18.6)

30. Secondary Outcome: Period 2: Cmax: Maximum Observed Plasma Total Radioactivity Concentration for [14C]-TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq/mL
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
ng eq/mL | 39.85 (33.6)

31. Secondary Outcome: Period 2: Tmax: Time to Reach the Maximum Plasma Total Radioactivity Concentration (Cmax) for [14C]-TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 22
Measure: Median (Full Range); unit: hr
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
hr | 0.758 [0.51 to 1.51]

32. Secondary Outcome: Period 2: AUCt: Area Under the Plasma Total Radioactivity Concentration-time Curve From Time 0 to Time of the Last Common Time Point t for [14C]-TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
ng eq*hr/mL | 109.0 (25.6)

33. Secondary Outcome: Period 2: AUClast: Area Under the Plasma Total Radioactivity Concentration-time Curve From Time 0 to Last Quantifiable Concentration for [14C]-TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
ng eq*hr/mL | 135.5 (20.2)

34. Secondary Outcome: Period 2: AUC∞: Area Under the Plasma Total Radioactivity Concentration-time Curve From Time 0 to Infinity for [14C]-TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: PK Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Participants who received the dose of [14C]-TAK-906 50 mg oral solution in Treatment Period 2 were evaluated for this outcome measure. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 5
ng eq*hr/mL | 144.3 (19.0)

35. Secondary Outcome: Period 2: t(1/2)z: Terminal Disposition Phase Half-life of Plasma Total Radioactivity Concentration for [14C]-TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose in Treatment Period 2
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 5
hr | 35.539 (26.2)

36. Secondary Outcome: Period 2: Cmax: Maximum Observed Whole Blood Total Radioactivity Concentration for [14C]-TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq/mL
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
ng eq/mL | 28.41 (26.7)

37. Secondary Outcome: Period 2: Tmax: Time to Reach the Maximum Whole Blood Total Radioactivity Concentration (Cmax) for [14C]-TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 2
Population: as for outcome 22
Measure: Median (Full Range); unit: hr
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
hr | 0.504 [0.50 to 1.50]

38. Secondary Outcome: Period 2: AUClast: Area Under the Whole Blood Total Radioactivity Concentration-time Curve From Time 0 to Last Quantifiable Concentration for [14C]-TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose in Treatment Period 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 6
ng eq*hr/mL | 83.17 (13.1)

39. Secondary Outcome: Period 2: AUC∞: Area Under the Whole Blood Total Radioactivity Concentration-time Curve From Time 0 to Infinity for [14C]-TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 2
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 5
ng eq*hr/mL | 87.25 (13.8)

40. Secondary Outcome: Period 2: t(1/2)z: Terminal Disposition Phase Half-life of Whole Blood Total Radioactivity Concentration for [14C]-TAK-906 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Treatment Period 2
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | [14C]-TAK-906 50 mg
Number analyzed (Participants) | 5
hr | 16.964 (112.1)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 ± 2 days after last dose of the study drug (Up to approximately 41 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Population included all participants who received at least one dose of the study drug. As prespecified in the protocol data for adverse events was collected and reported for Treatment Period 1 and Treatment Period 2.
Groups:
- TAK-906 50 mg + [14C]-TAK-906 100 μg: TAK-906 50 mg, capsule, orally, followed by [14C]-TAK-906 100 μg (approximately 1 μCi), infusion, intravenously, once on Day 1 of Treatment Period 1.
Arm/Group | TAK-906 50 mg + [14C]-TAK-906 100 μg | [14C]-TAK-906 50 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-906 50 mg + [14C]-TAK-906 100 μg (N=6) | [14C]-TAK-906 50 mg (N=6)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT04454918/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT04454918/SAP_001.pdf